CLINICAL TRIAL: NCT06219174
Title: Targeting ODC as an Immunotherapeutic Target in STK11 (LKB1) Pathway-Deficient NSCLC
Brief Title: Targeting ODC as an Immunotherapeutic Target in STK11 (LKB1) Pathway-Deficient NSCLC (DFMO)
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Drugs unavailable
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20386
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Non Small Cell Lung Cancer; Lung Cancer
Keywords: Pembrolizumab; Difluoromethylornithine
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — pembrolizumab; Eflornithine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1: Dose Escalation for Pembrolizumab and Difluoromethylornithine (DFMO) (Experimental): Difluoromethylornithine (DFMO) + Pembrolizumab Pre-treated or treatment naive advanced or metastatic NSCLC.
  The phase I dose escalation will include a fixed dose of Pembrolizumab IV every 3 weeks and escalating doses of DFMO (three dose levels) to determine the maximum tolerated dose (MTD) to be used in the phase II portion of the trial.
  DFMO level -1: Dose Level -1: 4500 mg/m2 by mouth (PO) once a day (QD).
  DFMO Level 1: (start): 6750 mg/m2 PO QD
  Dose Level 2: 9000 mg/m2 PO QD
  Interventions: Drug: Pembrolizumab; Drug: Difluoromethylornithine
- Phase II: Pembrolizumab and Difluoromethylornithine (DFMO) (Active Comparator): Difluoromethylornithine (DFMO) + Pembrolizumab
  Advanced/metastatic NSCLC who are immunotherapy naïve.
  Pembrolizumab IV flat dose every 3 weeks
  DFMO dose to be determined (TBD) based on maximum tolerated dose (MTD) and dose limiting toxicities (DLT) in Phase I dose escalation.
  Interventions: Drug: Pembrolizumab; Drug: Difluoromethylornithine

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg IV Q3 weeks
  Other Names: Keytruda
Drug: Difluoromethylornithine — Dose Level -1: 4500 mg/m2 by mouth (PO) daily Dose Level 1: 6750 mg/m2 by mouth (PO) daily Dose Level 2: 9000 mg/m2 by mouth (PO) daily
  Other Names: DFMO

SUMMARY:
The purpose of this study is to establish the safety, toxicity, and tolerability of Difluoromethylornithine (DFMO) in combination with pembrolizumab in advanced/metastatic Non-Small Cell Lung Cancer (NSCLC). Researchers also want to investigate how effective DFMO is at treating patients with advanced/ metastatic NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be willing and able to provide written informed consent/assent for the trial.
* Patients must be ≥ 18 years of age on day of signing informed consent.
* Patients must have measurable disease based on RECIST 1.1
* Patients must have archival tissue where available. Patients enrolled on the phase 1 escalation trial where archival tissue is not available will undergo a fresh biopsy where clinically feasible after discussion with the sponsor.
* Patients enrolled on the Phase II trial must be willing and able to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion.
* Tumor proportional score of PD-L1 ≥1%
* Patients must have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Patients must demonstrate adequate organ function on all screening labs. Screening labs should be performed within 10 days of treatment initiation.
* Histologically confirmed NSCLC that is at advanced/metastatic stage and for which there is no standard therapy option likely to convey clinical benefit. Advanced/metastatic is defined as unresectable or metastatic disease. Patients must have exhausted all approved available therapies.
* Patients must harbor an STK11 mutation via CLIA-certified assay.
* Phase I: Maybe treatment naïve or pretreated for advance or metastatic NSCLC. Patients whose tumors harbor an activating mutation (including but not limited to EGFR, ALK, ROS1) are eligible if they were previously treated with targeted therapy.
* Phase II: Patients must be treatment naïve in the stage IV setting, with the exception of patients whose tumors harbor an activating mutation (including but not limited to EGFR, ALK, ROS1) and were previously treated with targeted therapy.
* Female patients of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication.
* Female patients of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication.
* Male patients should agree to use an adequate method of barrier contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* Patients cannot have clinically significant hearing loss that requires a hearing aid.

Exclusion Criteria:

* Patients who are currently participating in and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Patients that have a diagnosis of immunodeficiency or is receiving systemic steroid therapy at doses ≥ 10 mg prednisone or any other form of systemic immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Patients that have a known history of TB Disease (Mycobacterium tuberculosis).
* Patients that have a hypersensitivity to pembrolizumab, DFMO or any of its excipients.
* Patients enrolled on the phase II trial, who have had prior treatment with a PD1 or PDL1 inhibitor, anti-CTLA 4 antibody or any other antibody or drug that specifically targets immune checkpoint pathway in the stage IV setting (i.e. not "immune therapy naïve").
* Patients who have received thoracic radiation >30Gy within six months of the first dose of pembrolizumab.
* Patients that had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Patients that have received major surgery must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Patients that have a known additional malignancy that is progressing or requires active treatment.

Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer.

* Patients that have a known active central nervous system (CNS) metastasis and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they have stable CNS disease for at least 4 weeks prior to enrollment, have known treated and asymptomatic brain metastases and not using steroids in doses greater than 10 mg of prednisone daily (or equivalent). This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Patients that have active autoimmune disease that has required systemic treatment in the past 2 years.
* Patients that have an active infection requiring systemic therapy.
* Patients that have a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, that would substantially increase risk of incurring adverse events (AEs) from the study medications, that would interfere with the subject's participation for the full duration of the trial or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Patients that have a known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the trial.
* Patients that have a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Patients that have known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Patients that have received a live vaccine within 30 days of planned start of study therapy.
* Patients that have a history of, or any evidence of active non-infectious pneumonitis that required or requires steriods.
* Patients that have evidence of interstitial lung disease (ILD).
* Patients that have a history of symptomatic (NYHA class II-IV) heart failure.
* Patients harboring STK11 variants listed in ClinVAR as benign or likely-benign will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Phase I- Maximum Tolerated Dose (MTD) | Up to 12 Months
  To determine the maximum tolerated dose (MTD) and recommended phase II dose (R2PD) of DFMO in combination with pembrolizumab. The MTD will be declared if 1 or fewer patients have a Dose limiting toxicity (DLT) in that dose level.
Phase II- Objective Response Rate (ORR) | Up to 5 Years
  To determine the efficacy of DFMO in combination with pembrolizumab. Objective response is defined as confirmed complete response (CR) or confirmed partial response (PR) based on modified RECIST guidelines version 1.1.

SECONDARY OUTCOMES:
Phase II- Progression Free Survival (PFS) | Up to 5 Years
  Progression-free survival will be measured from the start of treatment with pembrolizumab and DFMO until the documentation of disease progression or death due to any cause, whichever occurs first. For subjects who are alive and progression-free at the time of data cut-off for analysis, PFS will be censored at the last tumor assessment date.
Phase II- Overall Survival (OS) | Up to 5 Years
  Overall survival will be determined as the time from the start of treatment with pembrolizumab and DFMO until death due to any cause. For subjects who are alive at the time of data cut-off, OS will be censored on the last date when subjects are known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Jhanelle E. Gray, M.D., Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center's Clinical Trials Website — http://www.moffitt.org/clinicaltrials